CLINICAL TRIAL: NCT01863004
Title: Proteasomal Inhibition for Patients With Mis-sense Mutated Dysferlin
Acronym: Dysferlin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient enrollment rate
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DYSF001A1; 2011DR1148 (Registry Identifier: Swissmedic Referenznummer 2011DR1148)
Record Dates: First submitted 2013-04-29; First posted 2013-05-27 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Dysferlinopathy
MeSH Terms: conditions — Dysferlinopathy | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Velcade®) (Experimental): This study tests whether salvage of mis-sense mutated dysferlin through proteasomal inhibition seen in cultured muscle cells can be translated into patients harboring dysferlin mis-sense mutations. The proteasomal inhibitor Bortezomib (Velcade®) is already approved as a medication for the treatment of multiple myeloma in Switzerland and in other countries.
  Following an administration of a single dose of Bortezomib repeated needle muscle biopsies and blood draws will be performed to assess dysferlin levels in skeletal muscle and blood monocytes over a five day period.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib
  Other Names: Velcade®

SUMMARY:
Dysferlin is a protein with an important role in the repair of muscle surface membranes. Mutations in dysferlin cause different forms of muscular dystrophies. Dysferlinopathies are inherited in an autosomal recessive manner, and many patients with this disease harbor mis-sense mutations in at least one of their two pathogenic DYSF alleles. These patients have significantly reduced or absent dysferlin levels in skeletal muscle, suggesting that dysferlin encoded by mis-sense alleles is rapidly degraded by the cell's quality-control system. In a series of in-vitro experiments we showed that mis-sense mutated dysferlin can be salvaged from degradation by proteasomal inhibition. This resulted in an increase of functional dysferlin protein and a subsequent repair of plasma membranes of cultured patient-derived muscle cells. In this proof-of-concept study we would like to test wether proteasomal inhibition can salvage mis-sense mutated dysferlin in patients harboring certain dysferlin mis-sense mutations.

ELIGIBILITY:
Inclusion Criteria:

* must carry at least one allele of a salvageable mis-sense mutation of dysferlin
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Bleeding disorder
* Acute or chronic kidney failure (CCL <50 ml/min)
* Advanced liver disease or active hepatitis
* Congestive heart failure NYHA III and IV
* Pregnancy or nursing
* Immunosuppression (prednisolone doses below 20 mg/d are allowed)
* Therapy with strong inhibitors of cytochrome P450 3A4
* HCV or HIV infection
* Regular alcohol consumption (>14 drinks a week)
* Drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-12; Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Dysferlin protein expression levels change from baseline over 5 days assessed by repeated biopsies and blood draws in skeletal muscle and in blood monocytes following administration of a single dose of Bortezomib. | repeated needle muscle biopsies over a five day period
  Repeated needle muscle biopsies and blood draws will be performed after administration of a single dose of Bortezomib (Velcade) to assess dysferlin protein expression in skeletal muscle and in blood monocytes over a five day period.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sinnreich, Prof. Dr. MD, Principal Investigator — Sponsor-Investigator, Neuromuscular Center, Neurology Clinic, University Hospital Basel, Switzerland
Locations (1):
- Neuromuskuläres Zentrum, Universitätsspital Basel, Basel, Switzerland

REFERENCES:
- [Result] Azakir BA, Di Fulvio S, Kinter J, Sinnreich M. Proteasomal inhibition restores biological function of mis-sense mutated dysferlin in patient-derived muscle cells. J Biol Chem. 2012 Mar 23;287(13):10344-10354. doi: 10.1074/jbc.M111.329078. Epub 2012 Feb 8. PMID 22318734 (Retraction: PMID 28754767 J Biol Chem. 2017 Jul 28;292(30):12542)
- [Result] Di Fulvio S, Azakir BA, Therrien C, Sinnreich M. Dysferlin interacts with histone deacetylase 6 and increases alpha-tubulin acetylation. PLoS One. 2011;6(12):e28563. doi: 10.1371/journal.pone.0028563. Epub 2011 Dec 8. PMID 22174839 (Retraction: PMID 29377932 PLoS One. 2018 Jan 29;13(1):e0192239)
- [Result] Azakir BA, Di Fulvio S, Salomon S, Brockhoff M, Therrien C, Sinnreich M. Modular dispensability of dysferlin C2 domains reveals rational design for mini-dysferlin molecules. J Biol Chem. 2012 Aug 10;287(33):27629-36. doi: 10.1074/jbc.M112.391722. Epub 2012 Jun 26. PMID 22736764 (Retraction: PMID 28754768 J Biol Chem. 2017 Jul 28;292(30):12543)